CLINICAL TRIAL: NCT02894060
Title: A Study of Immunological Biomarkers as Predictors of Cardiovascular Events
Acronym: BIOKID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PI2013_843_0019
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Cardiovascular Abnormalities
Keywords: Cardiovascular events
MeSH Terms: conditions — Cardiovascular Abnormalities | interventions — Hematologic Tests

ARMS (1):
- blood (Experimental): blood tests
  Interventions: Other: blood tests

INTERVENTIONS:
Other: blood tests — Blood tests done by the nurse in the CRC (clinical research center). The quantity of blood taken wil be (3 5-mL tubes):
  2 plain tubes and 1EDTA tube Arterial blood pressure will be measured at the CRC. Then, an X-ray of the profile of the abdomen will be taken without preparation to evaluate aortic calcification (in the radiology department of the Amiens hospital)

SUMMARY:
Cardiovascular disease linked to atherosclerosis (e.g. infarcts, cerebro-vascular accidents) are one of the main causes of mortality in the general population. The recruitment of macrophages from the walls of the arterial lumen followed by unregulated capture of oxidated LDL (LDLox) leads to the accumulation of cholesterol esters and the formation of foamy cells characteristic of fatty streaks, the first phase of atherogenesis. These fatty streaks are rarely followed by clinical events, but can progress to complicated atheromatoses (calcification, rupture) resulting in the occurrence of various clinical events such as myocardial infarction and cerebro-vascular accidents (CVA). Once oxidated, LDL becomes immunogenic and induces anti-LDLox antibody production that could be markers of progression of atherosclerosis. During LDL oxidation, a multitude of specific oxidative epitopes (SOE) such as oxidated phospholipids (PLox) and malondialdehyde-lysine epitopes (MDA) are generated. In order to measure the level of markers in the blood, researchers developed a series of immunologic levels in vitro, using specific antibodies directed against well-defined epitopes. Recently, it was shown that Lp(a ) would be the preferred transporter of these PLox. In fact, several clinical studies show a strong correlation between PLox/apoB concentrations and Lp(a). This marker (PLox/apoB) predicts future morbidity and mortality due to cardiovascular diseases, including CVA, up to 15 years in advance, independent of all other known risk factors. CD36 is a scavenger receptor that recognizes LDLox, but more specifically PLox present in these lipoproteins .One soluble form of inflammatory CD36 (sCD36) was recently identified. In this study, only healthy volunteers were recruited in order to be able to establish normal serum ranges of different immunologic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Persons providing signed informed consent
* Persons with healthcare coverage

Exclusion Criteria:

* Renal disease
* Cardiovascular disease
* Auto immune disease
* Pregnancy in progress
* Infection
* Dementia
* Persons under legal protection
* Malnutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Blood level of immunologic biomarker PLox/apoB | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Michel ANDREJAK, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France